CLINICAL TRIAL: NCT04511091
Title: Studio Osservazionale Retrospettivo Uneventful Vatslobectomy: Caratteristiche Cliniche
Brief Title: Studio Osservazionale Retrospettivo Uneventful Vatslobectomy: Caratteristiche Cliniche All'Interno Del Registro Vats Group
Acronym: VATS
Status: Completed | Type: Observational
Sponsor: University Hospital of Ferrara (Other)
Responsible Party: Principal Investigator, Pio Maniscalco, Medical Doctor, Thoracic Surgeon, University Hospital of Ferrara
Other Study IDs: EM352-2020_AOUFe/171173_EM1
Record Dates: First submitted 2020-08-10; First posted 2020-08-12 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Thoracic Surgery, Video-Assisted
Keywords: VATS; lobectomy; length-of-stay; hospitalization; fast-track; discharge

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Vats Group: patients underwent planned VATS lobectomy for NSCLC from the Italian VATS Group Database (a validated, risk-adjusted, prospective, outcomes-based program with 50 participating hospitals in Italy) were included in the analysis.
  Interventions: Procedure: VATS lobectomy

INTERVENTIONS:
Procedure: VATS lobectomy — VATS lobectomy allows surgeons to carry out exactly the same operation within the chest that is performed by thoracotomy, but it is done through 3-4 small incisions without rib spreading rather than the large incision with rib spreading that a thoracotomy entails. The surgeon gains his view inside the chest from a small video camera inserted through one of the small incisions, and the procedure is carried out with long instruments passed through the other small incisions.

SUMMARY:
Background VATS lobectomy centers face pressure to reduce hospitalization to contain costs, and some centers have sought to develop "fast-track" protocols. There are limited data to identify which patients would be appropriate for fast-tracking.

Objective The first objective was to identify factors associated to short lenght of stay after VATS lobectomy. The second objective was to verify the influence of these variables in uncomplicated VATS lobectomy.

Methods We reviewed all thoracoscopic lobectomies for cancer operations reported to the Italian VATS Group between January 2014 and January 2020. Patient and procedural characteristics, length of stay and 30-day morbidity and mortality were reviewed. Patients were divided into two subgroups depending on their reaching the targeted length of stay (≤ or > 4 days). The association between preoperative and intraoperative variables and postoperative length of stay (LOS) ≤ 4 days was assessed using a stepwise multivariate logistic regression analysis to identify factors independently associated with LOS and factors related to LOS in uncomplicated cases.

DETAILED DESCRIPTION:
Data source The Italian VATS Group Database is a validated, risk-adjusted, prospective, outcomes-based program with 50 participating hospitals in Italy. The VATS Group Database collects data on different variables on a standardized data form: patient demographics informations, surgical interventions, medical history, cancer staging and outcome. Patients' outcomes are reviewed and records are updated the first time at 30 days after surgery, then at 180 days. Next update is recorded at 6 months from surgery and every 6 months for the first 2 years of follow-up, and annually thereafter. The VATS Group Database implements rigorous quality assurance and safety procedures to maintain a high level of accuracy and security of data.

The study has been approved by hospital ethics committee. The current analysis was reviewed and approved for scientific merit and feasibility by the VATS Group Scientific Committee and presented at the annual VATS Group meeting.

Patient population and study design Study population consisted of patients who received intended VATS lobectomy as the primary procedure for NSCLC at VATS Group participating centres and included in the VATS Group database between January 2014 and January 2020. We excluded all patients with incomplete clinical, intraoperative and postoperative data. Data entered from centers sporadically (less than 10 cases per year) were also excluded.

In order to analyse the factors related to lenght of stay, the study design provides a comparison between two groups of patients: the first group, identified as "LOS ≤ 4" including all patient disharged within 4 days after surgery, while the second group, called "LOS > 4" including all cases discharged after the fourth postoperative day.

Covariates We compared selected clinical variables to analyse the presence of a possible association with lenght of stay: data were divided into preoperative, intraoperative and postoperative.

Furthermore, three groups were made according to the number of cases entered by the different centers and considered as a possible influential variable: group A (less than 50 cases), group B (number of cases between 51 and 100) and group C (above 100 patients).

Statistical Analysis Patient baseline demographic and comorbidity variables were analyzed using frequencies and proportions for categorical variables and means, standard deviations (SDs), medians and interquartile ranges (IQR) for continuous variables.

The comparisons between groups (LOS ≤ 4 vs LOS > 4) categories were made by the following tests: Student t-test for continuous variables with approximately normal distribution, non-parametric Wilcoxon Mann Whitney test for other numerical variables and for categorical variables Pearson's chi-square test or Fisher's exact test in the case of low-volume categories were adopted.

To investigate the factors independently associated with the hospital stay outcome we used simple logistic regression models with the variables of interest, and a simplified multiple model with a stepwise backward procedure to obtain a more parsimonious model that contained only the significant factors. Covariates of interest were patients' demographics, co- morbidities, hospital lobectomy volume , operative features, pain relief techniques, type of surcial approach. A significance level of 0.2 was required to enter the model and a level of 0.05 was required to remain in the model. Adjusted odds ratios (ORs) and 95% confidence intervals (95% CIs) were presented. All P-values are two sided with statistical significance evaluated at the 0.05 α level. All tests were performed with Stata 13.0 statistical software (Stata Corp, College Station, TX).

ELIGIBILITY:
Inclusion Criteria:

* Patients of the Italian VATS Group Database between January 2014 and January 2020

Exclusion Criteria:

* Patients not included in the Italian VATS Group Database;
* all patients with incomplete clinical, intraoperative and postoperative data and data entered from centers sporadically (less than 10 cases per year) were also excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients were divided into two subgroups depending on their reaching the targeted length of stay (≤ or > 4 days). The association between preoperative and intraoperative variables and postoperative length of stay (LOS) ≤ 4 days was assessed using a stepwise multivariate logistic regression analysis to identify factors independently associated with LOS and factors related to LOS in uncomplicated cases.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
to identify factors associated to short lenght of stay after VATS lobectomy | 2014-2020
  to identify factors associated to short lenght of stay after VATS lobectomy

SECONDARY OUTCOMES:
to verify the influence of these variables (factors associated to short lenght of stay) in uncomplicated VATS lobectomy | 2014-2020
  to verify the influence of these variables (factors associated to short lenght of stay) in uncomplicated VATS lobectomy

CONTACTS AND LOCATIONS:
Overall Officials: GIORGIO CAVALLESCO, Professor, Study Director — Università degli Studi di Ferrara

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Romano PHP, Ritley D. Selecting Quality and Resource Use Measures: A Decision Guide for Community Quality Collaboratives. Agency for Healthcare Research and Quality, Rockville, MD 2010 pp. 1-106.
- [Background] Carey K. Measuring the hospital length of stay/readmission cost trade-off under a bundled payment mechanism. Health Econ. 2015 Jul;24(7):790-802. doi: 10.1002/hec.3061. Epub 2014 May 7. PMID 24803387
- [Background] Osnabrugge RL, Speir AM, Head SJ, Jones PG, Ailawadi G, Fonner CE, Fonner E Jr, Kappetein AP, Rich JB. Prediction of costs and length of stay in coronary artery bypass grafting. Ann Thorac Surg. 2014 Oct;98(4):1286-93. doi: 10.1016/j.athoracsur.2014.05.073. Epub 2014 Aug 7. PMID 25110338
- [Background] Wright CD, Gaissert HA, Grab JD, O'Brien SM, Peterson ED, Allen MS. Predictors of prolonged length of stay after lobectomy for lung cancer: a Society of Thoracic Surgeons General Thoracic Surgery Database risk-adjustment model. Ann Thorac Surg. 2008 Jun;85(6):1857-65; discussion 1865. doi: 10.1016/j.athoracsur.2008.03.024. PMID 18498784
- [Background] Farjah F, Lou F, Rusch VW, Rizk NP. The quality metric prolonged length of stay misses clinically important adverse events. Ann Thorac Surg. 2012 Sep;94(3):881-7; discussion 887-8. doi: 10.1016/j.athoracsur.2012.04.082. Epub 2012 Jun 27. PMID 22742847
- [Background] Cattaneo SM, Park BJ, Wilton AS, Seshan VE, Bains MS, Downey RJ, Flores RM, Rizk N, Rusch VW. Use of video-assisted thoracic surgery for lobectomy in the elderly results in fewer complications. Ann Thorac Surg. 2008 Jan;85(1):231-5; discussion 235-6. doi: 10.1016/j.athoracsur.2007.07.080. PMID 18154816
- [Background] Francis N, Kennedy RH, Ljungqvist O, Mythen MG. Manual of fast track recovery for colorectal surgery. Berlin: Springer; 2012.
- [Background] Gimenez-Mila M, Klein AA, Martinez G. Design and implementation of an enhanced recovery program in thoracic surgery. J Thorac Dis. 2016 Feb;8(Suppl 1):S37-45. doi: 10.3978/j.issn.2072-1439.2015.10.71. PMID 26941969
- [Background] Gonfiotti A, Viggiano D, Voltolini L, Bertani A, Bertolaccini L, Crisci R, Droghetti A. Enhanced recovery after surgery and video-assisted thoracic surgery lobectomy: the Italian VATS Group surgical protocol. J Thorac Dis. 2018 Mar;10(Suppl 4):S564-S570. doi: 10.21037/jtd.2018.01.157. PMID 29629203
- [Background] Paton F, Chambers D, Wilson P, Eastwood A, Craig D, Fox D, Jayne D, McGinnes E. Effectiveness and implementation of enhanced recovery after surgery programmes: a rapid evidence synthesis. BMJ Open. 2014 Jul 22;4(7):e005015. doi: 10.1136/bmjopen-2014-005015. PMID 25052168
- [Background] Giambrone GP, Smith MC, Wu X, Gaber-Baylis LK, Bhat AU, Zabih R, Altorki NK, Fleischut PM, Stiles BM. Variability in length of stay after uncomplicated pulmonary lobectomy: is length of stay a quality metric or a patient metric?dagger. Eur J Cardiothorac Surg. 2016 Apr;49(4):e65-71. doi: 10.1093/ejcts/ezv476. Epub 2016 Jan 27. PMID 26823164
- [Background] Paul S, Sedrakyan A, Chiu YL, Nasar A, Port JL, Lee PC, Stiles BM, Altorki NK. Outcomes after lobectomy using thoracoscopy vs thoracotomy: a comparative effectiveness analysis utilizing the Nationwide Inpatient Sample database. Eur J Cardiothorac Surg. 2013 Apr;43(4):813-7. doi: 10.1093/ejcts/ezs428. Epub 2012 Jul 22. PMID 22826474
- [Background] Mathisen DJ. Re: Video-assisted thoracoscopic surgery versus open lobectomy for primary non-small-cell lung cancer: a propensity-matched analysis of outcome from the European Society of Thoracic Surgeon database. Eur J Cardiothorac Surg. 2016 Feb;49(2):609-10. doi: 10.1093/ejcts/ezv167. Epub 2015 Apr 28. No abstract available. PMID 25920462
- [Background] Berrisford R, Brunelli A, Rocco G, Treasure T, Utley M; Audit and guidelines committee of the European Society of Thoracic Surgeons; European Association of Cardiothoracic Surgeons. The European Thoracic Surgery Database project: modelling the risk of in-hospital death following lung resection. Eur J Cardiothorac Surg. 2005 Aug;28(2):306-11. doi: 10.1016/j.ejcts.2005.03.047. PMID 16144067
- [Background] Sanchez-Lorente D, Navarro-Ripoll R, Guzman R, Moises J, Gimeno E, Boada M, Molins L. Prehabilitation in thoracic surgery. J Thorac Dis. 2018 Aug;10(Suppl 22):S2593-S2600. doi: 10.21037/jtd.2018.08.18. PMID 30345096
- [Background] Augustin F, Maier HT, Weissenbacher A, Ng C, Lucciarini P, Ofner D, Ulmer H, Schmid T. Causes, predictors and consequences of conversion from VATS to open lung lobectomy. Surg Endosc. 2016 Jun;30(6):2415-21. doi: 10.1007/s00464-015-4492-3. Epub 2015 Sep 3. PMID 26335073
- [Background] Park JS, Kim HK, Choi YS, Kim J, Shim YM, Kim K. Unplanned conversion to thoracotomy during video-assisted thoracic surgery lobectomy does not compromise the surgical outcome. World J Surg. 2011 Mar;35(3):590-5. doi: 10.1007/s00268-010-0913-6. PMID 21181470
- [Background] Decaluwe H, Petersen RH, Hansen H, Piwkowski C, Augustin F, Brunelli A, Schmid T, Papagiannopoulos K, Moons J, Gossot D; ESTS Minimally Invasive Thoracic Surgery Interest Group (MITIG). Major intraoperative complications during video-assisted thoracoscopic anatomical lung resections: an intention-to-treat analysis. Eur J Cardiothorac Surg. 2015 Oct;48(4):588-98; discussion 599. doi: 10.1093/ejcts/ezv287. PMID 26385060
- [Background] Harris CG, James RS, Tian DH, Yan TD, Doyle MP, Gonzalez-Rivas D, Cao C. Systematic review and meta-analysis of uniportal versus multiportal video-assisted thoracoscopic lobectomy for lung cancer. Ann Cardiothorac Surg. 2016 Mar;5(2):76-84. doi: 10.21037/acs.2016.03.17. PMID 27134832
- [Background] Maggino L, Liu JB, Ecker BL, Pitt HA, Vollmer CM Jr. Impact of Operative Time on Outcomes after Pancreatic Resection: A Risk-Adjusted Analysis Using the American College of Surgeons NSQIP Database. J Am Coll Surg. 2018 May;226(5):844-857.e3. doi: 10.1016/j.jamcollsurg.2018.01.004. Epub 2018 Mar 1. PMID 29408353
- [Background] Magee MJ, Herbert MA, Tumey L, Prince SL. Establishing a Dedicated General Thoracic Surgery Subspecialty Program Improves Lung Cancer Outcomes. Ann Thorac Surg. 2017 Apr;103(4):1063-1069. doi: 10.1016/j.athoracsur.2016.09.033. Epub 2016 Dec 8. PMID 27938908
- [Background] Park HS, Detterbeck FC, Boffa DJ, Kim AW. Impact of hospital volume of thoracoscopic lobectomy on primary lung cancer outcomes. Ann Thorac Surg. 2012 Feb;93(2):372-9. doi: 10.1016/j.athoracsur.2011.06.054. Epub 2011 Sep 25. PMID 21945225
- [Background] Otake H, Yasunaga H, Horiguchi H, Matsutani N, Matsuda S, Ohe K. Impact of hospital volume on chest tube duration, length of stay, and mortality after lobectomy. Ann Thorac Surg. 2011 Sep;92(3):1069-74. doi: 10.1016/j.athoracsur.2011.04.087. PMID 21871302
- [Background] Kamiyoshihara M, Nagashima T, Ibe T, Atsumi J, Shimizu K, Takeyoshi I. Is epidural analgesia necessary after video-assisted thoracoscopic lobectomy? Asian Cardiovasc Thorac Ann. 2010 Oct;18(5):464-8. doi: 10.1177/0218492310381817. PMID 20947601
- [Background] Piccioni F, Ragazzi R. Anesthesia and analgesia: how does the role of anesthetists changes in the ERAS program for VATS lobectomy. J Vis Surg. 2018 Jan 11;4:9. doi: 10.21037/jovs.2017.12.11. eCollection 2018. PMID 29445595
- [Background] Daly DJ, Myles PS. Update on the role of paravertebral blocks for thoracic surgery: are they worth it? Curr Opin Anaesthesiol. 2009 Feb;22(1):38-43. doi: 10.1097/ACO.0b013e32831a4074. PMID 19237975